CLINICAL TRIAL: NCT06679400
Title: Effects of Myofascial Massage and Patient-therapist Communication Levels on Shoulder Muscle Properties in Breast Cancer Survivors With Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, David B Lipps, PhD, Associate Professor of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00250137; U24AT011969 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Pain, Myofacial
Keywords: Massage therapy; Ultrasound; History of unilateral breast cancer
MeSH Terms: conditions — Facial Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to receive massage where communication with the massage therapist is permitted or restricted.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Massage with communication level 1 (Experimental): The therapist and the participant will have this level of communication (known as level 1 here). Further details will be explained at the end of the study.
  Interventions: Behavioral: Massage
- Massage with communication level 2 (Experimental): The therapist and the participant will have this level of communication (known as level 2). Further details will be explained at the end of the study.
  Interventions: Behavioral: Massage

INTERVENTIONS:
Behavioral: Massage — Participants will have one massage that will last 30 minutes and focus on the chest and shoulder of the side that received the cancer treatment. There will be certain techniques applied during the intervention (per protocol). The timing and order of each element will be varied based on tissue response and patient feedback.
  All participants will have ultrasounds and complete surveys prior and after the massage.

SUMMARY:
The objective of the proposed study is to assess how myofascial massage alters stiffness and microvascular perfusion of shoulder muscles and how these changes are influenced by patient-therapist interactions.

The primary hypothesis is that stiffness of shoulder muscles will be decreased, and microvascular perfusion will be increased after a 30-minute myofascial massage, and that the addition of patient-therapist communication levels will result in greater changes with certain levels.

DETAILED DESCRIPTION:
Please note that there are certain details left off of this registration in order to collect information regarding certain aspects of the trial. These details (approved by the IRB) will be updated at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Previous unilateral breast cancer diagnosis
* Treatment for primary breast cancer was completed 3 months to 2 years prior to enrollment (defined as completion of all treatments except oral maintenance therapies)
* Myofascial pain in upper quadrant of the chest
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Chronic neuromuscular or orthopedic injury currently affecting upper extremity function that is unrelated to their cancer diagnosis
* Currently undergoing physical therapy, occupational therapy or other treatment for side effects related to their cancer diagnosis or other injury to the upper extremity
* History of fibromyalgia
* Broken or bruised skin in the chest/shoulder area
* Diagnosed with metastatic breast cancer
* Currently receiving treatment for other forms of cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle stiffness of the pectoralis major | Baseline, post massage (approximately 30 minutes and 60 minutes)
  This will be assessed by ultrasound shear wave elastography before and after myofascial massage.

SECONDARY OUTCOMES:
Change in muscle perfusion of the pectoralis major and upper trapezius | Baseline, post massage (approximately 30 minutes and 60 minutes)
  This will be assessed by Doppler imaging and superb microvascular imaging before and after myofascial massage.
Change in muscle stiffness of the pectoralis major compared between groups | Baseline, post massage (approximately 30 minutes and 60 minutes)
  This will be assessed by ultrasound shear wave elastography and compared between patients randomized to a group with restricted or unrestricted communication with the massage therapist.
Global Satisfaction measured by the Patient Global Impression of Change will be compared between groups at the different communication levels | Approximately 60 minutes (during wait period after massage)
  This is a one question that participants chose from Very much improved (0) - Very much worse (6).

CONTACTS AND LOCATIONS:
Overall Officials: David Lipps, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT06679400/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT06679400/ICF_001.pdf